CLINICAL TRIAL: NCT04210154
Title: Comparison of Pre- and Post-dilution Hemodiafiltration Modalities - Effects on Biocompatibility and Solute Clearance in Children
Brief Title: Comparison of Pre- vs Post-dilution Haemodiafiltration in Children
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: Istanbul University (Other); Heidelberg University (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 19BO27
Record Dates: First submitted 2019-12-11; First posted 2019-12-24 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Haemodiafiltration
Keywords: Haemodiafiltration; Haemodialysis; Children
MeSH Terms: interventions — Hemodiafiltration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Haemodiafiltration — pre-dilution and post-dilution Haemodiafiltration

SUMMARY:
Cardiovascular morbidity and mortality are increased in children on conventional haemodialysis. Haemodiafiltration (HDF) is a newer type of dialysis which has two main types (post-dilution and predilution HDF). Post-dilution HDF is associated with better vascular health, blood pressure and growth in children. Furthermore, pre-dilution HDF is shown to remove a wider spectrum of uremic toxin compared to post-dilution HDF in adults. The investigators need more data to define the optimum dialysis modality for children.

DETAILED DESCRIPTION:
Hypothesis: In children with end stage kidney disease pre-dilution HDF (pre-HDF) achieves improved clearances across a wide molecular weight range compared to post-dilution HDF (post-HDF).

Plan of Investigation: Prevalent patients on thrice weekly HD or HDF who have a single pool Kt/v>1.2 will be randomized in to either study arm A (pre-HDF, post-HDF) or B (post-HDF, pre-HDF) after a conditioning period on post-HDF. Dialysis prescription will be kept constant during study periods including blood flow, dialysate flow, dialysate content, filter type and size. Pre-dialysis and post-dialysis bloods will be drawn at baseline and at the end of each treatment with either modality. Reduction ratios of small and middle molecular weight toxins and protein bound toxins as well as markers of inflammation and nutrition will be compared between two modalities. Assessment of blood pressure (ambulatory blood pressure monitoring) and patient wellbeing (questionnaire) will be performed at the end of each period.

Children will be recruited from paediatric dialysis units in London, Istanbul Heidelberg and Lyon with extension to other centres to be confirmed.

Outcomes: If the results of this study demonstrate better clearance with pre-dilution HDF compared to post-dilution HDF, this will inform a future long-term outcome study comparing different HDF modalities and will contribute to define optimum dialysis modality for children.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated in paediatric dialysis centres between 5-20 years of age
2. Receiving maintenance haemodialysis with HD or HDF for the preceding 3 months
3. In post-dilution HDF for at least 4 weeks before the start of the study
4. Patients with stable vascular access (central line or arteriovenous fistula) and no plan to change access modality for the duration of the study
5. Provision for ultrapure water for HDF (defined as containing <0.1 colony forming unit /ml and <0.03 endotoxin unit/ml) documented in the month prior to study start

Exclusion Criteria:

1. Incident dialysis patients (on HD or HDF for < 3 months)
2. Patients with acute infections in the preceding 2 weeks
3. Patients with underlying chronic inflammatory disorders (Including vasculitis)
4. Single pool Kt/V less than 1.2 in the month prior to the study start.
5. Children who have haemoglobin concentrations lower than 10 g/dL

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children on thrice weekly maintanenece HD or HDF
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Removal of middle molecular weight uremic toxins | 4 weeks
  The outcome measure is the difference in Beta2-microglobulin reduction ratios between pre- and post-dilution HDF treatments.

SECONDARY OUTCOMES:
Removal of low molecular weight | 4 weeks
  Comparison of urea and creatinine reduction ratios between pre- and post-dilution HDF modalities
Removal of protein bound uremic toxins | 4 weeks
  Comparison of indole acetate and p-cresyl sulphate reduction ratios between pre- and post-dilution HDF modalities
Comparison of biocompatibility by using an inflammation markers | 4 weeks
  Comparison of high sensitive C reactive protein, interleukin 6 and tumor necrosis factor alfa reduction ratios between pre- and post-dilution HDF modalities
Removal of nutritional markers | 4 weeks
  Comparison of Leptin and Ghrelin reduction ratios between pre- and post-dilution HDF modalities
Assessment of blood pressure by Ambulatory blood pressure monitoring (ABPM) | 4 weeks
  Comparison of systolic and diastolic blood pressures between pre- and post-dilution HDF modalities
Child Quality of Life (QoL) questionnaire | 4 weeks
  Questionnaire including information on post-dialysis recovery time, physical activity, school or college attendance and sleep pattern will be recorded by the patient. Questionnaire will be performed at the end of each period with pre- and post-dilution HDF modality. Scale 1 to 5 - higher scores indicate better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Rukshana Shroff, MD PhD, Study Chair — Great Ormond Street Children's Hospital, London, UK; Salim Caliskan, Prof Dr, Principal Investigator — Istanbul University, Cerrahpasa Medical Faculty, Istanbul, Turkey; Nur Canpolat, Assoc Prof, Principal Investigator — Istanbul University, Cerrahpasa Medical Faculty, Istanbul, Turkey; Ayse Agbas, MD, Principal Investigator — University of Health Sciences, Haseki Education and Research Hospital, Istanbul, Turkey
Locations (4):
- Division of Pediatric Nephrology Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Lyon, Bron, France
- Division of Pediatric Nephrology Center for Pediatrics and Adolescent Medicine, Heidelberg, Germany
- Istanbul University-Cerrahpasa, Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)
- Great Ormond Street Children's Hospital, London, United Kingdom